CLINICAL TRIAL: NCT01107288
Title: A Randomized Controlled Trial of Music-Based Multitask Exercises (Jaques-Dalcroze Eurhythmics) on Gait, Balance and Fall Risk in the Elderly
Brief Title: Effects of a Music-Based Multitask Exercises Program on Gait, Balance and Fall Risk in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Jaques-Dalcroze Institute, Geneva, Switzerland (Unknown)
Responsible Party: Principal Investigator, Andrea Trombetti, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 07-156
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Gait; Balance; Falls
Keywords: Aged; Balance; Dual-task; Exercise; Falls; Gait; Music
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Randomized to receive the intervention first
  Interventions: Other: Music-based multitask exercises program
- Delayed intervention control group (Other): Randomized to wait-list control first
  Interventions: Other: Music-based multitask exercises program

INTERVENTIONS:
Other: Music-based multitask exercises program — Subjects are entered into a 6-month Jaques-Dalcroze eurhythmics program and are followed for an additional 6 months after the intervention period. They complete assessments at baseline, 6 and 12 months. The program consists of structured 1-hour group exercises classes, conducted weekly by an experimented instructor, that include varied multitask exercises performed to the rhythm of improvised piano music, sometimes with the manipulation of objects (e.g., instruments of percussion, balls), with gradually increasing difficulty over time. Basic exercises consist of walking following the music, responding directly to changes in music's rhythmic patterns.
  Other Names: Jaques-Dalcroze Eurhythmics
  Arms: Intervention group
Other: Music-based multitask exercises program — Subjects are wait-listed to receive, 6 months after randomization, the same 6-month Jaques-Dalcroze eurhythmics program as the Intervention group. They complete assessments at baseline, 6 and 12 months.
  Other Names: Jaques-Dalcroze Eurhythmics
  Arms: Delayed intervention control group

SUMMARY:
The aim of this study is to investigate the effectiveness of a 6-month music-based multitask exercises program (Jaques-Dalcroze eurhythmics) in improving gait and balance, and reducing fall risk in community-dwelling older adults with an increased risk of falling.

DETAILED DESCRIPTION:
Background

Falls are among the most common and devastating concern facing older adults. The scope of this problem will continue to expand as the number of older adults is projected to increase dramatically over the coming decades. Since most falls occur as a result of a complex interaction of risk factors, considerable evidence documents that gait instability and poor balance capacity are two major contributors to falling. A large proportion of falls in elderly people are experienced while walking and, with advancing age, older adults are more likely to fall when they are engaged in concurrent tasks. Gait variability, particularly during dual-task walking conditions, may provide an objective measure to characterize impaired execution of gait, with greater variability placing older adults at increased risk of falling.

Jaques-Dalcroze eurhythmics, an approach to music education through movement developed by the composer Emile Jaques-Dalcroze (1865-1960) in Geneva in the early 20th century, is currently practiced worldwide in the field of music, as well as dance, theatre and therapy. Initially intended for music students, Jaques-Dalcroze eurhythmics soon expanded extensively to music education of children and adolescents all over the world. The main focus of this method are on developing rhythmicality and musicality as well as strengthening body awareness, coordination, expression, as verbal and social skills. Recently, Jaques-Dalcroze eurhythmics classes for older adults were developed. Those classes engage the elderly in varied multitask exercises performed to the rhythm of improvised piano music, sometimes with the manipulation of objects (e.g., instruments of percussion, balls). Basic exercises consist of walking following the music, responding directly to changes in music's rhythmic patterns. In a cross-sectional study performed in long-term Jaques-Dalcroze eurhythmics users, the age-related increase of stride-to-stride variability appeared to be attenuated (Kressig, 2005). The effectiveness of this intervention to achieve improvement in gait variability in older adults without previous experience of Jaques-Dalcroze eurhythmics need to be confirmed prospectively.

Method

This randomized controlled trial was designed to assess the efficacy of a 6-month community-based Jaques-Dalcroze eurhythmics program in improving gait and balance, and reducing fall risk in elderly people with an increased risk of falling. The primary objective is to assess the efficacy of the intervention in reducing gait variability. Change in gait variability under dual-task condition over 6 months is the primary endpoint. The main secondary objectives are to assess the effects on other quantitative gait and balance measures, functional tests performances, and falls.

Volunteer participants are recruited in the Geneva area (Switzerland) through flyers, press releases and advertisements in local community newspapers. Individuals aged 65 or older, community-dwelling and identified at high risk for falling are randomly assigned, according to a computer-generated list, to either an immediate Jaques-Dalcroze eurhythmics program of weekly 1-hour classes for 6 months or a wait-list control group scheduled to receive the same intervention 6 months following the completion of the baseline assessment. Participants in the intervention group are followed for an additional 6 months in order to evaluate whether intervention gains can be maintained over time. Main outcome measures include gait (under single and dual-task conditions) and balance performances assessed by quantitative analysis (i.e., electronic walkway and angular velocity transducers) and functional tests administered at baseline, 6 and 12 months. Falls data are prospectively ascertained during the whole follow-up using a monthly calendar method with daily records. The principal analysis will be done on an intention to treat basis.

Following completion of the 12-month follow-up, subjects will have the option of continuing classes via the Jaques-Dalcroze Institute. Subjects will be invited to enter into an extension phase of the trial and participate in a follow-up assessment visit scheduled four years following original trial enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Living in the community
* Without previous Jaques-Dalcroze eurhythmics experience (except during childhood)
* Identified as being at high risk of fall (i.e., one or more self-reported falls after the age of 65 years or balance impairment as assessed by a simplified Tinetti test higher than 2 over 7 or the presence of one or two indicators of physical frailty based on Fried's criteria)

Exclusion Criteria:

* Neurological or orthopaedic disease (e.g., stroke with residual motor deficit, Parkinson's disease, osteoarthritis) with a significant impact on gait and balance performances
* Progressive or unstable medical conditions that could limit participation (e.g., terminal illness)
* Fully dependent on an assistive device such as canes and walkers

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in gait variability | 6 months

SECONDARY OUTCOMES:
Change in other spatio-temporal gait parameters | 6 months, 12 months
Change in balance measures (Trunk sway parameters) | 6 months, 12 months
Change in functional tests performances (Timed Up & Go test and simplified Tinetti test) | 6 months, 12 months
Number of falls, fallers and multiple fallers (Daily recording of falls using falls calendars, to be returned monthly) | 6 months, 12 months
Change in quality of life (SF-12 Health Survey questionnaire), anxiety/depression (HAD scale), cognitive function (Mini-Mental State Examination, Frontal Assessment Battery, clock drawing test), nutritional status (Mini Nutritional Assessment tool) | 6 months, 12 months
Change in gait variability | 12 months
Change in all outcome measures | 4 years
  Long-term extension study

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Trombetti, MD, Principal Investigator — Bone Diseases Service, Department of Rehabilitation and Geriatrics, University Hospitals and Faculty of Medicine of Geneva
Locations (1):
- Department of Rehabilitation and Geriatrics, Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Trombetti A, Hars M, Herrmann FR, Kressig RW, Ferrari S, Rizzoli R. Effect of music-based multitask training on gait, balance, and fall risk in elderly people: a randomized controlled trial. Arch Intern Med. 2011 Mar 28;171(6):525-33. doi: 10.1001/archinternmed.2010.446. Epub 2010 Nov 22. PMID 21098340